CLINICAL TRIAL: NCT04663880
Title: Validation Study of the ALYATEC Allergen Exposure Chamber by Determining the Concentration of House Dust Mite Allergen Inducing Early and/or Late Bronchial Response in Asthmatic Subjects Allergic to Mite
Brief Title: Validation of Strasbourg Environmental Exposure Chamber ALYATEC in Mite Allergic Subjects With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ALY-001
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Allergic Asthma; Allergy to House Dust; Allergy
Keywords: Allergy; Asthma; House dust mite
MeSH Terms: conditions — Hypersensitivity; Asthma

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, cross-over study including two study groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthmatic subjects allergic to house dust mite (Experimental): 24 subjects were randomized in a doubleblinded manner into six subgroups. All were exposed first to placebo then in cross over to three different Der p1 concentrations, respectively 15, 25, and 46 ng/m3.
  Interventions: Other: Exposure to placebo in EEC; Other: Exposure to three concentrations of HDM allergen in EEC
- Asthmatic subjects not allergic to house dust mite (Active Comparator): 13 subjects were exposed first to placebo then to Der p1 concentration of 25 ng/m3.
  Interventions: Other: Exposure to placebo in EEC; Other: Exposure to a single concentration of HDM allergen in EEC

INTERVENTIONS:
Other: Exposure to placebo in EEC — Patients are exposed to placebo (saline solution) in the EEC for 4h maximum
Other: Exposure to three concentrations of HDM allergen in EEC — Patients are exposed to different concentrations of airborne HDM allergen (Der p1) in the EEC for 4h maximum
  Arms: Asthmatic subjects allergic to house dust mite
Other: Exposure to a single concentration of HDM allergen in EEC — Patients are exposed to a single concentration of airborne HDM allergen (Der p1) in the EEC for 4h maximum
  Arms: Asthmatic subjects not allergic to house dust mite

SUMMARY:
This is a randomized, double blind, cross-over study designed to determine the concentration of airborne house dust mite allergen inducing bronchial response in asthmatic subjects allergic to mite, during allergen exposures in the Alyatec environmental exposure chamber (EEC).

The study was also designed to validate the specificity of the asthmatic reaction induced by exposure to airborne house dust mite allergen in Alyatec EEC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having signed the informed consent
* Subjects affiliated to a social security scheme
* Positive metacholine test
* FEV1 value > 70% of theoretical FEV1 value
* Asthma Control Test (ACT) ≥ 20/25 in 4 weeks prior to EEC exposure

Group A:

* Mild allergic asthma to HDM (GINA 1 or 2) with associated rhinitis and/or conjunctivitis.
* Positive skin prick-test to Dpt and Df (wheal diameter >5 mm compared to the negative control)
* Specific immunoglobulin E (IgE) for Dpt and Df > 0.7 kU/L

Group B:

* Mild allergic asthma (GINA 1 or 2) not sensitized to HDM with associated rhinitis and/or conjunctivitis.
* Negative skin prick-test and specific IgE for Dpt and Df.
* Positive skin prick-test and specific IgE for another allergen.

Exclusion Criteria:

* Uncontrolled asthma
* Asthma Control Test (ACT) < 20/25 in 4 weeks prior to EEC exposure
* Use of oral corticosteroids in the 4 weeks preceding inclusion in the study
* Use of biotherapy in the 4 months preceding inclusion in the study
* Existence of a severe obstructive syndrome with FEV1 <70% of the theoretical value
* Obstruction triggered by spirometric evaluations
* Hospitalization for asthma or exacerbation in the last 4 weeks
* History of Acute Severe Asthma requiring hospitalization in intensive care or intubation
* Desensitization to dust mite allergens in the last 5 years
* Sensitization to allergens in the indoor environment (cat allergens or molds) with obvious exposure to these allergens
* Active tobacco: plus 10 cigarettes / day and tobacco history of +10 PA
* Uncontrolled systemic arterial hypertension
* Recent myocardial infarction (<3 months)
* Recent stroke (<3 months)
* Known arterial aneurysm
* Epilepsy under treatment
* Progressive tumor pathology
* Chronic renal pathology
* Hypersensitivity to one of the excipients used
* Subjects who participated in another clinical study in the three months prior to inclusion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Determine the concentration of HDM allergen (in ng/m3 of Der p1) necessary to induce a bronchial response in at least 60% of asthmatic subjects allergic to HDM | 10 hours: 4 hours of exposure in the EEC then 6 hours post-exposure.
  The bronchial response is evaluated by measuring FEV1 value during EEC exposure.
  Early asthmatic response (EAR) occurs when a 20% drop in FEV1 is detected during the exposure compared to the pre-exposure FEV1.
  Late bronchial response (LAR) occurs when a 15% drop in FEV1 or 20% drop in peak flow is detected 1 to 6h after the EAR.

SECONDARY OUTCOMES:
Evaluate the safety of allergenic exposure in EEC | 28 hours: 4 hours of exposure in EEC then 24 hours post-exposure
  Safety is assessed with clinical evaluations performed during the 4h of exposure in the EEC
Evaluate the metrology of the EEC | 4 hours of exposure in EEC
  The metrology is assessed with the measure of allergen concentration and particules diameter thanks to sensors in the chamber.
Evaluate the specificity of the bronchial response | 4 hours of exposure in EEC
  The specificity of the bronchial response is assessed with the HDM exposure in the EEC of asthmatic subjects non allergic to HDM.
Evaluate the effect of the exposure on rhinitis symptoms | 28 hours: 4 hours of exposure in EEC then 24 hours post-exposure
  The effect of the exposure on the rhinitis response is assessed with Total Nasal Symptom Score (TNSS).
  The TNSS was obtained from the sum of all four individual symptom scores, with a total possible score ranging from 0 (no symptoms) to 12 (maximum symptom intensity).
Evaluate the effect of the exposure on conjunctivitis symptoms | 28 hours: 4 hours of exposure in EEC then 24 hours post-exposure
  The effect of the exposure on the conjunctivitis response is assessed with Total Ocular Symptom Score (TOSS).
  The TOSS was obtained from the sum of all four individual symptom scores, with a total possible score ranging from 0 (no symptoms) to 12 (maximum symptom intensity).

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric de Blay, Pr., Principal Investigator — Alyatec
Locations (1):
- Alyatec, Strasbourg, Grand Est, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khayath N, Doyen V, Gherasim A, Radu C, Choual I, Beck N, Jacob A, Schoettel F, Vecellio L, Domis N, de Blay F. Validation of Strasbourg environmental exposure chamber (EEC) ALYATEC(R) in mite allergic subjects with asthma. J Asthma. 2020 Feb;57(2):140-148. doi: 10.1080/02770903.2018.1563902. Epub 2019 Mar 28. PMID 30919704
- See also: Alyatec website — https://www.alyatec.com/en/